CLINICAL TRIAL: NCT03327597
Title: Iceland Screens, Treats or Prevents Multiple Myeloma
Acronym: iStopMM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: Landspitali University Hospital (Other); Union for International Cancer Control (Other); Icelandic Heart Association (Other); deCODE genetics (Industry); International Myeloma Foundation/Black Swan Research Initiative (Unknown); The Binding Site (Unknown); Memorial Sloan Kettering Cancer Center (Other); European Research Council (Other); The Icelandic Centre for Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: UI-2017-MGUS
Record Dates: First submitted 2017-10-19; First posted 2017-10-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance
Keywords: MGUS; Screening; Population-based
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance | interventions — Mental Health; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and participants will be blinded to what participants are in the normal group and which participants are in arm 1 in the MGUS-group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Abnormal Non-MGUS (Active Comparator): Participants previously diagnosed with MGUS, multiple myeloma or other lymphoproliferative disease.
  Interventions: Other: Mental Health and Quality of Life questionnaire; Other: Standard follow-up or treatment.
- MGUS group arm 1 (Experimental): Participants diagnosed with MGUS, randomized to group 1.
  Interventions: Other: Clinical follow-up 1; Other: Mental Health and Quality of Life questionnaire
- MGUS group arm 2 (Experimental): Participants diagnosed with MGUS, randomized to group 2.
  Interventions: Other: Mental Health and Quality of Life questionnaire; Other: Clinical follow-up 2
- MGUS group arm 3 (Experimental): Participants diagnosed with MGUS, randomized to group 3.
  Interventions: Other: Mental Health and Quality of Life questionnaire; Other: Clinical follow-up 3
- Normal group (Active Comparator): Participants without MGUS.
  Interventions: Other: Mental Health and Quality of Life questionnaire
- Controls (Active Comparator): Participants without MGUS, matched to MGUS participants by age and gender.
  Interventions: Other: Mental Health and Quality of Life questionnaire; Other: Clinical follow-up control

INTERVENTIONS:
Other: Clinical follow-up 1 — Participants receive routine care outside the bounds of the trial. No further work-up.
  Arms: MGUS group arm 1
Other: Mental Health and Quality of Life questionnaire — Participants receive a Mental Health and Quality of Life questionnaire that will be answered electronically on the study website (www.blodskimun.is)
Other: Standard follow-up or treatment. — Participants previously diagnosed as having MGUS or participants that have multiple myeloma or other lymphoproliferative diseases will receive standard clinical follow-up and treatment.
  Arms: Abnormal Non-MGUS
Other: Clinical follow-up 2 — Standard clinical follow-up according to International Myeloma Working Group (IMWG) guidelines.
  Arms: MGUS group arm 2
Other: Clinical follow-up 3 — Intensive clinical follow-up with regular clinical assessment, laboratory testing and radiology imaging.
  Arms: MGUS group arm 3
Other: Clinical follow-up control — Control clinical visit
  Arms: Controls

SUMMARY:
This study will assess the benefits and harms of screening for monoclonal gammopathy of undetermined significance (MGUS). The overall and disease-specific mortality will be compared between screened and not screened participants. All individuals registered as inhabitants in Iceland and born in 1975 or earlier have been invited to participate. The hypothesis is that an early detection of multiple myeloma (MM), through follow-up of MGUS, will improve overall survival and decrease complications associated with diagnosis and treatment of MM.

DETAILED DESCRIPTION:
Monoclonal gammopathy of undetermined significance (MGUS) is an asymptomatic premalignant stage that almost always precedes multiple myeloma (MM) and amyloidosis. It is defined by a monoclonal-(M)-protein detected on serum protein electrophoresis or immunofixation electrophoresis and can be diagnosed with a blood sample. Approximately four percent of individuals 50 years or older have MGUS which is associated with a 1-2% annual risk of malignant transformation but it is impossible to predict which individuals diagnosed as having MGUS will progress and receive a diagnosis of malignant disease.

To date, no evidence is available on the benefits and harms of population-based screening for MGUS and data from prospective studies that assess the optimal follow-up of MGUS are lacking.

All individuals that are registered as inhabitants in Iceland and born in 1975 or earlier have been invited to participate in the study. After signing informed consent, serum from the participants will be analysed for MGUS. The participants will not be contacted for blood sampling. Instead, an innovative approach will be used by taking advantage of the fact that most people 40 years or older do a blood test for various reasons during a three year period. The ID-list of participants in the study will be cross-linked with all major laboratories in Iceland, covering approximately 90% of all blood sampling in Iceland. When a participant has a blood test, a small amount (1 ml) of serum will be sampled and put in a separate test tube belonging to the study and used for diagnosis of MGUS.

Participants diagnosed as having MGUS will be randomized to three different arms, of which two arms will be called into a clinical study center for two separate types of follow-up. In arm one the participants will be asked to answer an electronic Mental Health and Quality of Life questionnaire annually but receive no active follow-up. In arm two and three the participants will be asked to answer the Mental Health and QoL questionnaire but also receive follow-up according to the International Myeloma Working Group (IMWG) guidelines (arm two) or intensive (arm three) clinical follow-up. Participants without MGUS will be asked to answer Mental Health and QoL questionnaire annually.

Results from two recent, population-based studies shows that early detection of MM through follow-up of MGUS is associated with fewer major complications and 13-14% better overall survival as compared to individuals presenting with MM without previous diagnosis of MGUS.

This study aims to assess the benefits and harms of population-based screening for MGUS by analyzing overall and disease specific survival, complications associated with screening and the effects screening has on mental health and quality of life. Furthermore, the aim of the study is to evaluate the optimal follow-up strategy of MGUS and the cost-effectiveness of screening for MGUS.

ELIGIBILITY:
Inclusion Criteria:

* Born 1975 or earlier
* With registered address in Iceland on November 1st 2016

Exclusion Criteria:

* Prior multiple myeloma
* Lymphoproliferative disease
* Amyloidosis
* M-protein >30 g/L or involved:uninvolved serum FLC ratio >100

Individuals with prior history of MGUS will be offered to be randomized into either moderate or intensive clinical follow-up (arms 2 or 3).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80761 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years from study start.
  Number of participants alive in each study arm

SECONDARY OUTCOMES:
Cause specific survival | 5 years from study start
  Survival among participants diagnosed with multiple myeloma, lymphoproliferative disease and amyloidosis.
Cost-effectiveness of screening for MGUS | 5 years from study start
  Will be calculated in collaboration with the Department of economy at the University of Iceland and will include standard estimates as deemed appropriate.
Global satisfaction with one´s life as assessed by the Satisfaction with life (SWLS) | 5 years from study start.
  Satisfaction with life scale (SWLS) is administered at baseline and during follow-up to assess global satisfaction with one's life according to the respondent ́s personal values and criteria, and therefore, is free of the researchers' personal values and criteria of specific areas of life deemed as important. SWLS is a five item self-report scale used to measure global life satisfaction. The items are scored on a 7-point scale, ranging from one (strongly disagree) to seven (strongly agree). A higher score reflects a greater satisfaction with life. Scores within 0-4 indicate minimal, 5-9 mild, 10-14 indicate moderate, 15-19 moderately, and 20-27 severe depressive symptoms. An optimal clinical cut off point for a Major Depressive Disorder (MDD) diagnosis is estimated to be a score of 12 or greater.
Happiness as assessed by the Single item measure for happiness | 5 years from study start
  The happiness question is administered at baseline and during follow-up to assess happiness. A single item measure for happiness is one question measure that assesses happiness in an individual's life. Happiness is estimated by an individual's response to the question: "By taking into account all aspects of your life, how happy do you consider yourself?" that is scored on a 10-point scale ranging from one (very unhappy) to ten (very happy). Higher scores indicate more happiness.
Resilience as assessed by The Connor-Davidson resilience scale (CD-RISC) | 5 years from study start
  The Connor-Davidson resilience scale (CD-RISC) is administered once during the study period to assess and control for resilience. The CD-RISC is a 10-item self-report measure (i.e., the short form of the questionnaire) assessing resilience in the past month. Each item is assessed on a five-point scale ranging from zero to four. Scores on each item are summed, and therefore, the total scores range from zero to 40. Higher scores indicate more resilience.
Social support as assessed by the Multidimensional scale of perceived social support (MSPSS) | 5 years from study start
  Multidimensional scale of perceived social support (MSPSS) is administered once during the study period to assess and control for social support. The MSPSS is a 12-item self-report questionnaire addressing relationships with family, friends, and significant other in the areas of social popularity, respect, and areas directly related to social support. Each item is assessed on a six-point scale ranging from one (Very strongly disagree) to seven (Very strongly agree). Score on each item is summed and averaged to both calculate the total scores and scale scores. Higher scores indicate more social support. Mean scores ranging from 1 to 2.9 can be considered low support, a score of 3 to 5 can be considered moderate support, and a score from 5.1 to 7 can be considered high support.
Adverse childhood experiences as assessed by the Adverse childhood experiences international questionnaire (ACE-IQ) | 5 years from study start
  Adverse childhood experiences international questionnaire (ACE-IQ) is administered once during the study period to assess and control for adverse events in childhood. The ACE-IQ is 43-item self-report measure assessing adverse childhood experiences. Questions cover family dysfunction, physical, sexual and emotional abuse and neglect by parents or caregivers, peer violence, witnessing community violence, and exposure to collective violence. Some items are yes or no questions, while other items are assessed on a five-point scale ranging from one (Always) to five (Never) or a four-point scale ranging from one (Many times) to four (Never).
Depressive symptoms as assessed by the Patient health questionnaire (PHQ-9) | 5 years from study start
  Patient health questionnaire (PHQ-9) is administered at baseline and during follow-up to assess depressive symptoms. The PHQ-9 is a nine item self-report questionnaire that measures frequency of depressive symptoms in the past two weeks. Each item is scored on a 4-point scale ranging from zero (none at all) to three (nearly every day). Therefore, overall scores range from zero to 27, with a higher score indicating more severe depressive symptoms. Scores between 0-4 indicate minimal depressive symptoms, 5-9 indicate mild depressive symptoms, 10-14 indicate moderate depressive symptoms, 15-19 indicate moderately severe depressive symptoms, and 20-27 indicate severe depressive. In addition, an optimal clinical cut off point for a MDD diagnosis is estimated to be a score of 12 or greater.
Anxiety symptoms as assessed by the Generalized anxiety disorder (GAD-7) | 5 years from study start
  Generalized anxiety disorder (GAD-7) is administered at baseline and during follow-up to assess anxiety symptoms. The GAD-7 is a self-report measure that assesses frequency of anxiety symptoms in the past two weeks, which in part correspond to the diagnostic criteria of generalized anxiety disorder in the DSM-IV. The questionnaire consists of seven items that assess how often in the past two weeks respondents experienced various symptoms of anxiety (e.g., feeling nervous, anxious or on edge). Each item is assessed on a 4-point scale that ranges from zero (not at all) to three (nearly every day). Total scores therefore range from zero to 21, with a higher score indicating more severe anxiety symptoms. Scores between 0-4 indicate minimal anxiety symptoms, 5-9 mild anxiety symptoms, 10-14 moderate anxiety symptoms, and 15-21 severe anxiety symptoms (Spitzer et al., 2006). In addition, an optimal clinical cut off point for a GAD diagnosis is estimated to be a score of 10 or greater
Worry as assessed by the Single item measure for worry | 5 years from study start
  The worry question is administered at baseline and during follow-up to assess worry thoughts. The single item measure for worry is a single item measure for health-related worry. Worry is estimated by an individual's response to the question: "How much do you worry about your health?" that is scored on a 10-point scale ranging from one (very little) to ten (very much). Higher scores indicate more worry.
Stress as assessed by the Perceived stress scale (PSS-10) | 5 years from study start
  Perceived stress scale (PSS-10) is administered during follow-up. The PSS-10 is a 10-item self-report measure on the degree in which life situations are appraised as stressful (i.e., unpredictable, uncontrollable, and overloading). PSS-10 is a 10-item self-report measure that assess the degree to which life situations were appraised as stressful in the past month, in particular how unpredictable, uncontrollable, and overloading individuals find their lives. Each item measures the frequency on a 5-point scale that ranges from 0 (never) to 4 (very often). The total score is calculated by reversing scores on four positively phrased items, and thereafter, summing the scores on each item. Total scores range from 0 to 40. Scores between 0-13 indicate low perceived stress, 14-26 moderate perceived stress, and 27-40 high perceived stress.
Post-traumatic stress symptoms as assessed by the Posttraumatic stress disorder checklist for DMS-5 (PCL-5) including the Life Events Checklist for DSM-5 (LEC-5) | 5 years from study start
  Posttraumatic stress disorder checklist for DMS-5 (PCL-5) including the Life Events Checklist for DSM-5 (LEC-5) is administered during follow-up. The PCL-5 is a 20-item self-report measure that assesses the severity of PTSD symptoms in the past month. Each item assesses a symptom of PTSD. The items on the PCL-5 measure how much an individual has been bothered by each symptom associated with a particular stressful event on a five-point scale ranging from zero (not at all) to four (extremely). Total scores range from 0-80 and higher scores indicate more severe symptoms of PTSD. According to previous studies a score of 33 or higher indicates the presence of clinically significant PTSD symptoms. The LEC is a self-report instrument that screens for 16 lifetime traumatic events that are known to potentially result in clinically significant distress including PTSD, in addition, other stressful events not captured by the 16 items can be reported
Health as assessed by the 36-Item short form survey (SF-36) | 5 years from study start
  36-Item short form survey (SF-36) is administered during follow-up. The SF-36 is a 36-item questionnaire assessing physical functioning, bodily pain, role limitations due to physical health and personal or emotional problems, general psychiatric health, social functioning, energy and fatigue, and general health perceptions. The measure also includes a single item that provides an indication of perceived change in health. Each item is assessed on a six-point scale ranging from one to six, which are recoded per a scoring key so that values range from zero to 100. Scores indicate the percentage of total possible score achieved. All items are recoded so that a high score indicates a more favorable health state. Thereafter, the average score is calculated for each scale. Items that are left blank (missing data) are not considered when calculating the scale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sigurdur Y Kristinsson, Professor, Principal Investigator — University of Iceland
Locations (1):
- University of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eythorsson E, Rognvaldsson S, Thorsteinsdottir S, Einarsson Long T, Reed ER, Sigurdardottir GA, Vidarsson B, Onundarson PT, Agnarsson BA, Sigurdardottir M, Olafsson I, Thorsteinsdottir I, Sveinsdottir SV, Sigurdsson F, Thordardottir AR, Palsson R, Indridason OS, Jonsson A, Gislason GK, Olafsson A, Sigurdsson J, Steingrimsdottir H, Hultcrantz M, Durie BGM, Harding S, Landgren O, Aspelund T, Love TJ, Kristinsson SY. Development of a Multivariable Model to Predict the Need for Bone Marrow Sampling in Persons With Monoclonal Gammopathy of Undetermined Significance : A Cohort Study Nested in a Clinical Trial. Ann Intern Med. 2024 Apr;177(4):449-457. doi: 10.7326/M23-2540. Epub 2024 Apr 2. PMID 38560901
- [Derived] Sigurbergsdottir AY, Rognvaldsson S, Thorsteinsdottir S, Sverrisdottir I, Sigurethardottir GA, Vietharsson B, Onundarson PT, Agnarsson BA, Sigurethardottir M, Thornorsteinsdottir I, Olafsson I, Thornorethardottir AR, Gislason GK, Olafsson A, Hultcrantz M, Durie BGM, Harding S, Landgren O, Love TJ, Kristinsson SY. Disease associations with monoclonal gammopathy of undetermined significance can only be evaluated using screened cohorts: results from the population-based iStopMM study. Haematologica. 2023 Dec 1;108(12):3392-3398. doi: 10.3324/haematol.2023.283191. PMID 37439374
- [Derived] Thorsteinsdottir S, Gislason GK, Aspelund T, Rognvaldsson S, Oskarsson JThorn, Sigurethardottir GA, Thornorethardottir AR, Vietharsson B, Onundarson PT, Agnarsson BA, Sigurethardottir M, Thornorsteinsdottir I, Olafsson I, Eythornorsson E, Jonsson A, Berlanga O, Hultcrantz M, Durie BGM, Love TJ, Harding S, Landgren O, Kristinsson SY. Prevalence of smoldering multiple myeloma based on nationwide screening. Nat Med. 2023 Feb;29(2):467-472. doi: 10.1038/s41591-022-02183-6. Epub 2023 Feb 6. PMID 36747117